CLINICAL TRIAL: NCT02041351
Title: Docetaxel in Patients With Metastatic Breast Cancer Who Have Been Heavily Pretreated, Including Prior Treatment With Paclitaxel or Docetaxel.
Brief Title: Biweekly Docetaxel in Patients With Metastatic Breast Cancer.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centro Universitario contra el Cáncer (Other)
Responsible Party: Principal Investigator, Jesus Livio Jimenez Santos, medical oncology resident, Centro Universitario contra el Cáncer
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ON13-004
Record Dates: First submitted 2014-01-18; First posted 2014-01-22 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Metastatic Breast Cancer
Keywords: metastatic breast cancer; taxanes; heavily pretreated
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- docetaxel (Experimental): measurement evaluation every 2 months tomography of all measurable lesions in millimeters, to assess response rate, partial and complete responses.
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Docetaxel — evaluate the activity of docetaxel on, metastatic lesions when measured after 4 cycles of chemotherapy
  Other Names: evaluating the response rate and progression-free interval

SUMMARY:
There is clinical benefit of docetaxel administered to patients who have progressed to 3 or more lines of chemotherapy including prior exposure to paclitaxel or docetaxel; using docetaxel in metastatic stage breast cancer previously exposed to taxanes equal therapeutic responses are obtained that it never received taxanes.

DETAILED DESCRIPTION:
Methodology:

Prospective non-randomized phase IIa. The selected patients with metastatic breast cancer heavily pretreated including those previously treated with taxanes, receive docetaxel administered at a dose of 45mg/m2 body surface every 2 weeks to assess the activity of this drug.

Variables:

Age. Menopausal status. Hormone receptor status. Overexpression of HER2 neu. Location of metastatic sites. Performance status (PS) 0-3. comorbidities.

Case management in the variables (patient subgroups )

The patients with HER 2 neu overexpression of anti -HER2 therapy will further chemotherapy with docetaxel.

The patients presenting with brain metastases may receive radiation therapy to the brain and then at the end of radiotherapy, start docetaxel.

Patients whose tumors express estrogen receptors and progesterone positive receive treatment with docetaxel:

Where there is visceral crisis and it is shown that they have already progressed to more than 2 lines of previously administered hormone treatment.

In no event cytotoxic chemotherapy with concurrent docetaxel was administered to an anti-estrogen drug.

And they can continue only when hormone therapy has achieved complete response measurable lesions with docetaxel and opt for a non-cytotoxic anti-estrogen therapy and when it came to presenting unacceptable toxicity with docetaxel.

Evaluations:

clinical assessment that will include physical examination and review of laboratory studies were carried out every 2 weeks before authorizing the housing management of a next cycle.

The objective assessment of tumor response was carried out by imaging studies (CT) by RECIST criteria after administration of the 4 criteria of cycles, a cycle is administered every 2 weeks with docetaxel at a dose of 45mg/m2.

Response Criteria

1. Response tumor shrinkage by royalty over 30%.
2. Greater than 1 cm in the size of tumor lesions decrease.
3. Disease-free survival
4. Progression-free survival.
5. Stable disease
6. Improved quality of life that is decreased bone pain, improvement of dyspnea.

ELIGIBILITY:
Inclusion Criteria: Women over 21 years of age diagnosed with breast cancer in clinical stage IV, who had received 3 or more lines of cytotoxic chemotherapy, which may have included paclitaxel or docetaxel, which have measurable or evaluable tumor activity in any distant organ and who are fully conscious and well oriented to permit informed consent.

Exclusion Criteria:

Male patients with metastatic breast cancer. Patients with grade 3 neuropathy by prior exposure to taxanes. Patients under 21 and over 85 years of age. Metastasis of one site in the central nervous system.

Ages: 21 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2013-11; Primary Completion 2014-01 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
disease free interval | 4 months
  more than 4 months free of clinically detectable cancer until recurrent cancer is diagnosed

SECONDARY OUTCOMES:
partial response | 2 months
  Decreases measurable tumor mass by 50% after treatment, With the report of Decreased size in millimeters of the original tumor.
rate response | 3 months
  percentage of patients who responded with a decrease greater than 40% of the lesions at the time of initiation of this treatment after 3 months of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jesús L Santos, doctor, Principal Investigator — Centro Universitario contra el Cáncer U.A.N.L.
Locations (2):
- Mexico (2):
  - Centro Universitario Contra El Cáncer, Monterrey, Nuevo León
  - Jesus Livio Jimenez Santos, Monterrey, Nuevo León